CLINICAL TRIAL: NCT00483691
Title: Growth and Development Longitudinal Follow-Up
Brief Title: Trial of Home Visitation Among Infants With Failure To Thrive
Acronym: FTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Maureen Black, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTT
Record Dates: First submitted 2007-06-05; First posted 2007-06-07 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Failure to Thrive
Keywords: Intervention; Home Visit; Growth; Child Development
MeSH Terms: conditions — Failure to Thrive | interventions — House Calls

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Home Visit — Homw visits scheduled weekly for one year.

SUMMARY:
1. Children in the home intervention group will have better growth (increase in weight and height) than children in the control group.
2. Children in the home intervention group will have better behavior than children in the control group.
3. Children in the home intervention group will have better academic performance than children in the control group.

DETAILED DESCRIPTION:
During the first years of life when energy needs are high, growth serves as an objective measure of children's well-being. Failure-to-thrive (FTT) occurs when infants' rate of weight gain is below expectations based on age and gender-specific growth charts. The proposed randomized controlled trial evaluates whether a home-based intervention delivered by community health workers is effective in altering patterns of children's growth and development.

Infants were recruited from pediatric primary care clinics serving low-income, urban communities from 1988 through 1993. Eligibility criteria included age < 25 months, at least 35 weeks gestational age and appropriate birth weight for gestational age, and no congenital problems, disabilities, or chronic illnesses.

Children in the FTT group had to meet one of two criteria using age and gender-specific National Center for Health Statistics (NCHS) growth charts: sustained weight-for-age below the 5th percentile, weight-for-length below the 10th percentile or weight for age crossing two major centiles and falling below the 25th percentile. All infants were examined by a pediatrician, who also reviewed their medical charts to ensure that they met criteria for FTT and there were no known syndromes or obvious major organ system dysfunctions, such as congenital heart disease, to account for the growth failure of the infants in the FTT group.

Caregivers were invited to participate in a longitudinal research project, using consent procedures approved by the Institutional Review Board of the University of Maryland, Baltimore. Over 90% of eligible caregivers agreed and participated in an initial evaluation that included measures of growth, standardized developmental assessments, and a 60-minute interview of questionnaires on demographics, children's behavior, and maternal and family functioning. Developmental assessments were administered by psychology graduate students, supervised by a pediatric psychologist. A home visit was scheduled within two weeks of the initial evaluation.

Children with FTT were treated in an interdisciplinary clinic. Based on a randomization procedure, stratified by race, gender, and infant age to ensure equivalence across groups, children with FTT were randomized to receive either the clinical intervention plus home intervention (FTT-HI) or the clinical intervention only (FTT-CO).

The intervention was based on ecological theory and included a therapeutic alliance between the interventionist and the caregiver; support to the caregiver's personal, family, and environmental needs; opportunities to model and promote responsive parent-infant interaction; and problem-solving strategies regarding personal, parenting, and children's issues. The Hawaii Early Learning Program was used as a curriculum guide.

The intervention was delivered by three, part-time lay home visitors employed by a community-based agency specializing in early intervention. The home visitors received an eight-session training program and were supervised by a community health nurse. The home visitors had portable mats and toys to demonstrate developmentally appropriate activities and to facilitate parent-child interaction. They did not focus on nutrition or feeding behavior and they did not weigh the children. One-hour visits were scheduled weekly for one year; the number of visits varied from 0 to 47.

The children and caregivers return for regularly scheduled evaluations throughout the child's life. Evaluators are unaware of their growth or intervention status. Caregivers provide the name of the children's school and requests are sent for information on classroom behavior. Families and teachers are compensated for participating in evaluations.

The outcome measures are growth, cognition, academic performance, and social behavior. Evaluators are unaware of the children's growth history or group assignment. Standardized measures are used.

ELIGIBILITY:
Inclusion Criteria:

* Age < 25 months, at least 35 weeks gestational age, birth weight appropriate for gestational age, current weight-for-age < 5th percentile or weight-for-length < 10th percentile or weight for age crossing two major centiles and falling below the 25th percentile.

Exclusion Criteria:

* No congenital problems or developmental disabilities.

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 1989-01; Primary Completion 1995-12 (Actual); Study Completion 1995-12 (Actual)

PRIMARY OUTCOMES:
Growth, behavior, academic performance | 20 years
Growth | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Maureen M Black, Ph.D., Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland Growth and Nutrition Clinic, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Participants have been enrolled into a study funded by the Office of Child Abuse and Neglect with Dr. Dubowitz as PI.

REFERENCES:
- [Background] Black MM, Dubowitz H, Krishnakumar A, Starr RH Jr. Early intervention and recovery among children with failure to thrive: follow-up at age 8. Pediatrics. 2007 Jul;120(1):59-69. doi: 10.1542/peds.2006-1657. PMID 17606562
- [Result] Black MM, Dubowitz H, Hutcheson J, Berenson-Howard J, Starr RH Jr. A randomized clinical trial of home intervention for children with failure to thrive. Pediatrics. 1995 Jun;95(6):807-14. PMID 7539121